CLINICAL TRIAL: NCT07295665
Title: External Validation of Ischemia and Hemorrhage Risk Models in Patients With Coronary Heart Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xue Yu, Director of the Department of Cardiology, Beijing Hospital
Other Study IDs: 2025ZD0546402; 2025ZD0546402 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ischemic risk and bleeding risk model — This study verifies the ischemic risk and bleeding risk model developed in Project 1, compares the efficacy improvement of the new model with the traditional risk model, and verifies the effectiveness and stability of the model in different subgroups of the population, and assesses the generalizability of the model in real-world clinical practice, providing high-quality evidence-based basis for the formulation of individualized and precise antithrombotic strategies for coronary heart disease.

SUMMARY:
Thrombosis formation is the core mechanism for the occurrence of major adverse cardiovascular and cerebrovascular events in patients with coronary heart disease. Antithrombotic therapy is one of the most important treatment methods for secondary prevention of coronary heart disease. Antithrombotic drugs, while reducing ischemic events, often significantly increase the risk of bleeding. How to balance the risk of recurrent ischemic events and bleeding events in patients with coronary heart disease is a major challenge in the treatment of coronary heart disease. This project establishes a high-quality multicenter, prospective coronary heart disease cohort, with patients covering various clinical characteristics such as different regions, ages, and comorbidities. It verifies the ischemic risk and bleeding risk model developed in Project 1, compares the efficacy improvement of the new model with the traditional risk model, and verifies the effectiveness and stability of the model in different subgroups of the population, and assesses the generalizability of the model in real-world clinical practice, providing high-quality evidence-based basis for the formulation of individualized and precise antithrombotic strategies for coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Patients with clinically diagnosed various types of coronary heart disease, who are scheduled to receive long-term antithrombotic treatment;
* Patients with acute coronary syndrome or those who have undergone coronary intervention therapy, whose condition must be stable after treatment and meet the discharge criterias;

Exclusion Criteria:

* Combination of severe non-cardiovascular diseases: Expected lifespan does not exceed 6 months, such as patients with advanced cancer or other terminal diseases;
* Unable to cooperate with long-term follow-up: Such as patients with severe cognitive impairment or severe mental illness;
* Non-cardiovascular death within 24 hours after admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with clinically diagnosed various types of coronary heart disease, who are scheduled to receive long-term antithrombotic treatment;
  * Patients with acute coronary syndrome or those who have undergone coronary intervention therapy, whose condition must be stable after treatment and meet the discharge criterias;
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint | One year
  The primary efficacy endpoint is the major cardiovascular and cerebrovascular ischemic event (MACCE) during the 1-year follow-up period, which includes all-cause mortality, non-fatal myocardial infarction, unplanned revascularization, and stroke.
The primary safety endpoint | One year
  The primary safety endpoint is the major bleeding event (BARC type 3 and 5) during the 1-year follow-up period.